CLINICAL TRIAL: NCT03980210
Title: Effect of Hyperbaric Oxygen Therapy on Healthy Volunteers Microcirculation
Brief Title: Effect of Hyperbaric Oxygen Therapy on Microcirculation
Acronym: MICROHB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2018_63; 2019-A00053-54 (Registry Identifier: ID-RCB - ANSM)
Record Dates: First submitted 2019-05-15; First posted 2019-06-10 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Hyperbaric Oxygen Therapy
Keywords: Hyperbaric oxygen therapy; Normobaric oxygen therapy; Hyperoxia; Sidestream dark field videomicroscopy; Microcirculation
MeSH Terms: conditions — Hyperoxia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperbaric oxygen therapy (Experimental): Successive changes in fraction of inspired oxygen and barometric pressure (ATA: Atmosphere absolute)
  Five successive steps:
  1. FiO2 0.21 - 1 ATA
  2. FiO2 1 - 1 ATA
  3. FiO2 1 - 2.5 ATA
  4. FiO2 0.21 - 2.5 ATA
  5. FiO2 0.21 - 1 ATA
  Interventions: Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Procedure: Hyperbaric oxygen therapy — 1. FiO2 0.21 - 1 ATA
  2. FiO2 1 - 1 ATA
  3. FiO2 1 - 2.5 ATA
  4. FiO2 0.21 - 2.5 ATA
  5. FiO2 0.21 - 1 ATA

SUMMARY:
Previous studies shoes that hyperoxia alters microcirculation.The investigators hypothesize that hyperbaric may restore microcirculation integrity. This hypothesis is supported by a recent study in rabbits, but no data exists for humans.

The study will expose fifteen healthy volunteers to a succession of different fraction of inspired oxygen and barometric pressure and assess microcirculatory and macrocirculatory changes via sidestream dark field videomicroscopy, near-infrared spectroscopy, Laser Doppler, transthoracic echocardiography and bio-impedancemetry at every step.

DETAILED DESCRIPTION:
Microcirculation alterations and hyperoxia are known to alter ICU-patients' prognostic.

Studies have shown that hyperoxia alters healthy volunteers' microcirculation, whereas hyperbaric oxygen therapy is commonly used to facilitate cicatrization. There seems to be a paradox. A recent study in rabbits has given some evidences that hyperbaria may restore microcirculation integrity, but to date, there is no such evidences in human.

To study hyperoxia and hyperbaric induced changes in micro and macrocirculation, fifteen healthy volunteers will be exposed to successive variations of inspired oxygen fraction and barometric pressure according to a predefine sequence so that only one parameter will change from a condition to the next one :

1. FiO2 0.21 - 1 ATA
2. FiO2 1 - 1 ATA
3. FiO2 1 - 2.5 ATA
4. FiO2 0.21 - 2.5 ATA
5. FiO2 0.21 - 1 ATA

At each time, and after a 30 minutes period of exposure, measures will be made using SDF-microscopy, Laser Doppler and NIRS to assess microcirculation.

As previously described, macrocirculation can modify microcirculation due to a mechanism called hemodynamic coherence.

Hence, the investigators planned to assess macrocirculation changes at every step of the protocol using bioimpedancemetry and transthoracic echocardiography.

Each volunteer will be his own control, using the first measurements (condition 1. FiO2 0.21 - 1 ATA) as reference.

ELIGIBILITY:
Inclusion Criteria:

* To provide a medical certificate of fitness to dive (< 1 year)
* Consent given for study participation
* French health insurance affiliated

Exclusion Criteria:

* Temporary or definitive contra-indication to dive
* Pregnancy or < 18 years of age
* Precedent dive < 24 hours
* Under a legal protection measure
* Medical history of a disease known to alter microcirculation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-06-14 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Changes in proportion of perfused vessel (PPV) | 30 minutes after hyperbaric hyperoxia exposure (FiO2 1 - 2.5 ATA)
  Proportion of perfused vessel assessed by Sidestream dark field microscopy on the sublingual mucosa

SECONDARY OUTCOMES:
Changes in proportion of perfused vessel (PPV) | 30 minutes after FiO2 1 - 1 ATA exposure
  Proportion of perfused vessel assessed by Sidestream dark field microscopy on the sublingual mucosa
Changes in proportion of perfused vessel (PPV) | 30 minutes after FiO2 0.21 - 2.5 ATA exposure
  Proportion of perfused vessel assessed by Sidestream dark field microscopy on the sublingual mucosa
Changes in hyperemic reaction after a vaso-occlusion test | 30 minutes after FiO2 1 - 2.5 ATA exposure
  Area under curve assessed by near-infrared spectroscopy
Changes in area of hyperaemia after a vaso-occlusion test | 30 minutes after FiO2 1 - 2.5 ATA exposure
  Area under curve assessed by Laser-Doppler
Validation of cardiac output assessed by bioimpedancemetry under hyperbaric condition | 30 minutes after FiO2 1 - 2.5 ATA exposure
  Comparison with transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Thibault Duburcq, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHU, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cousin N, Goutay J, Girardie P, Favory R, Drumez E, Mathieu D, Poissy J, Parmentier E, Duburcq T. Effects of high oxygen tension on healthy volunteer microcirculation. Diving Hyperb Med. 2022 Dec 20;52(4):260-70. doi: 10.28920/dhm52.4.260-270. PMID 36525683